CLINICAL TRIAL: NCT02303483
Title: The Effect of Nicotinamide Ribose (NR) on Substrate Metabolism, Insulin Sensitivity, and Body Composition in Obese Men - a Randomized, Placebo Controlled Clinical Trial
Brief Title: The Effect of Vitamin B3 on Substrate Metabolism, Insulin Sensitivity, and Body Composition in Obese Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ole Dollerup, MD, PhD-student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 44081
Record Dates: First submitted 2014-11-20; First posted 2014-12-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Obese
MeSH Terms: conditions — Obesity | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): lime tablets
  Interventions: Dietary Supplement: Placebo
- Nicotinamide riboside (NR, Vit B3) (Experimental): NIAGEN (ChromaDex) 1 g x 2 orally per day
  Interventions: Dietary Supplement: Nicotinamide riboside (NIAGEN TM, ChromaDex, CA, USA )

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside (NIAGEN TM, ChromaDex, CA, USA )
  Arms: Nicotinamide riboside (NR, Vit B3)
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In animals, treatment with vitamin B3 improved insulin sensitivity and substrate metabolism. It is currently not know if vitamin B3 has the same positive effects in humans. In the current study the effect of a 3 month treatment with vitamin B3 on insulin sensitivity and substrate metabolism in obese men will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* written signed consent
* male
* BMI>30 kg/(m2)
* age: 40-70
* no medication
* non-smoker

Exclusion Criteria:

* endocrine disease
* other severe disease
* high daily activity level (>30 min / day)

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Change from baseline in insulin sensitivity at 3 months
  determined by a hyperinsulineamic clamp

SECONDARY OUTCOMES:
Substrate metabolism | Change from baseline in substrate metabolism at 3 months
  measured by indirect calorimetry
body composition | Change from baseline in body composition at 3 months
  measured by DEXA scan
Activation of satellite cells | Change from baseline in activation of satellite cells at 3 months
  measured by immunohistochemestry
lipid accumulation in liver and skeletal muscle tissue | Change from baseline in liver and muscle lipid content at 3 months
  determined by MR-spectroscopy
glucose turnover | Change from baseline in glucose turnover at 3 months
  determined by glucose tracer techniques
insulin signalling in skeletal muscle and adipose tissue biopsies | Change from baseline in insulin signaling at 3 months
  western blotting
Palmitate turnover | Change from baseline in palmitate turnover at 3 months
  determined by palmitate tracer techniques
Gut microbiota | Change from baseline in composition of gut microbiota at 3 months
  Intestinal bacteria composition by whole genome sequencing
Incretin hormone secretion | Change from baseline in incretion hormone secretion at 3 months
  Determined by measurement of incretin homones during an oral glucose tolerance test (OGTT)

CONTACTS AND LOCATIONS:
Overall Officials: Ole Dollerup, MD, Principal Investigator — The Novo Nordisk Foundation Center for Basic Metabolic Research, Integrative Physiology, University of Copenhagen
Locations (1):
- Medical Research Laboratories, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Dollerup OL, Chubanava S, Agerholm M, Sondergard SD, Altintas A, Moller AB, Hoyer KF, Ringgaard S, Stodkilde-Jorgensen H, Lavery GG, Barres R, Larsen S, Prats C, Jessen N, Treebak JT. Nicotinamide riboside does not alter mitochondrial respiration, content or morphology in skeletal muscle from obese and insulin-resistant men. J Physiol. 2020 Feb;598(4):731-754. doi: 10.1113/JP278752. Epub 2019 Dec 26. PMID 31710095
- [Derived] Dollerup OL, Trammell SAJ, Hartmann B, Holst JJ, Christensen B, Moller N, Gillum MP, Treebak JT, Jessen N. Effects of Nicotinamide Riboside on Endocrine Pancreatic Function and Incretin Hormones in Nondiabetic Men With Obesity. J Clin Endocrinol Metab. 2019 Nov 1;104(11):5703-5714. doi: 10.1210/jc.2019-01081. PMID 31390002
- [Derived] Dollerup OL, Christensen B, Svart M, Schmidt MS, Sulek K, Ringgaard S, Stodkilde-Jorgensen H, Moller N, Brenner C, Treebak JT, Jessen N. A randomized placebo-controlled clinical trial of nicotinamide riboside in obese men: safety, insulin-sensitivity, and lipid-mobilizing effects. Am J Clin Nutr. 2018 Aug 1;108(2):343-353. doi: 10.1093/ajcn/nqy132. PMID 29992272